CLINICAL TRIAL: NCT02366871
Title: The Safety of Oral Apixaban (Eliquis) Versus Subcutaneous Enoxaparin (Lovenox) for Thromboprophylaxis in Women With Suspected Pelvic Malignancy; a Prospective Randomized Open Blinded End-point (PROBE) Design
Brief Title: Oral Apixaban (Eliquis) Versus Enoxaparin (Lovenox) for Thromboprophylaxis in Women With Suspected Pelvic Malignancy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 15-0187.cc
Record Dates: First submitted 2015-02-02; First posted 2015-02-19 (Estimated); Results first posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Gynecologic Cancer; Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — apixaban; Enoxaparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral apixaban (Experimental): Oral apixaban 2.5 mg tablet twice daily for 28 days post-surgery
  Interventions: Drug: Oral apixaban
- Subcutaneous enoxaparin (Active Comparator): Subcutaneous enoxaparin 40mg once daily (QD) for 28 days post-surgery.
  Interventions: Drug: Subcutaneous enoxaparin

INTERVENTIONS:
Drug: Oral apixaban — To evaluate the incidence of major bleeding (including CRNM bleeding) events in women undergoing surgery for gynecologic cancer with apixaban 2.5 mg BID compared to current standard of care, subcutaneous enoxaparin 40 mg QD for 28 days post surgery.
  Other Names: Eliquis
  Arms: Oral apixaban
Drug: Subcutaneous enoxaparin — To evaluate the incidence of major bleeding (including CRNM bleeding) events in women undergoing surgery for gynecologic cancer with apixaban 2.5 mg BID compared to current standard of care, subcutaneous enoxaparin 40 mg QD for 28 days post surgery.
  Other Names: Lovenox
  Arms: Subcutaneous enoxaparin

SUMMARY:
The study will evaluate the incidence of major bleeding (including clinically relevant non-major (CRNM) bleeding) events in women undergoing surgery for gynecologic cancer with apixaban 2.5 mg twice a day (BID) compared to current standard of care, subcutaneous enoxaparin 40 mg once a day (QD) for 28 days post surgery.

DETAILED DESCRIPTION:
Apixaban (Eliquis) is an oral anticoagulant for the treatment and prevention of thromboembolic events. It is advantageous as there is no need to perform routine blood monitoring tests including, international normalized ratio (INR), partial thromboplastin time (PTT) and Factor Xa, to determine clotting in participants receiving treatment. Several studies have shown the efficacy of apixaban for the treatment and prevention of a venous thromboembolism (VTE).

We anticipate that the same efficacy could be replicated in the prevention of VTE in women undergoing surgery for gynecologic cancer. An oral-anticoagulant for standard treatment for prevention of VTE outcomes following surgery could help improve the surgical mortalities associated with gynecologic oncology surgical patients, improve patient adherence for outpatient treatment, and reduce VTE surveillance and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Suitable candidate for surgery (meets appropriate performance status, no significant cardiac/renal/hepatic dysfunction
* Diagnosis of pelvic malignancy (suspected/confirmed ovarian, endometrial/uterine, cervical cancers, and vulvar cancers) undergoing surgical debulking,
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to surgery,
* Women must not be breastfeeding, WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) apixaban plus 5 half-lives of study drug apixaban (2.5 days) plus 30 days (duration of ovulatory cycle) for a total of 32.5 days post-treatment completion.

Exclusion Criteria:

* Malignancy or mass that is non-gynecologic in origin (mass/tumor of origin other than reproductive organ such as rectal, abdominal, breast)
* Positive pregnancy test on day of surgery,
* Known history of Venous (Thromboembolism) VTE prior to diagnosis (DVT or Pulmonary Embolism (PE)) due to increased underlying risk of new event
* Concomitant NSAIDS or other anticoagulant/antiplatelet therapy including Acetylsalicylic Acid (Aspirin) (ASA) >81mg/day,
* Selective serotonin re uptake inhibitor (SSRIs) and Serotonin-nor-epinephrine re uptake inhibitor (SNRIs) (common anti-depressant therapies),
* Uncontrolled severe hypertension (systolic >200 mmHg or diastolic >120 mmHg),
* With prosthetic heart valves,
* Active bleeding condition (not limited to: thrombocytopenia, haemophilias, potential bleeding lesions, recent trauma or surgery, recent stroke, confirmed intracranial or intraspinal bleeding),
* Known or documented bleeding disorders not limited to: anti-phospholipid syndrome, homozygotes for Factor V Leiden deficiency, antithrombin III deficiency, protein C deficiency, Protein S deficiency, hyperhomocysteinemia, systemic lupus erythematous, or Prothrombin G2020 gene mutation,
* Significant renal disease as defined by creatinine clearance less than 30 mL/min,
* Significant liver disease as defined as Aspartate Transaminase (AST) or Alanine Transaminase (ALT) twice than normal,
* Concomitant use of dual strong inhibitors or inducers (CYP3A4, P-gp)
* Protein C deficiency (increased risk of skin necrosis do those on injectable anticoagulation),
* Documented allergy to apixaban and/or enoxaparin,
* Patient's deemed otherwise clinically unfit for clinical trial per Investigator's discretion

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saketh Guntupalli, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Southern California Keck School of Medicine, Los Angeles, California
  - University of Colorado Denver, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ross ME, Glickman A, Brennecke A, Tayebnejad A, Guntupalli SR. Adherence to postoperative thromboprophylactic medication among gynecologic oncology patients: A subanalysis. Gynecol Oncol. 2020 Sep;158(3):754-759. doi: 10.1016/j.ygyno.2020.06.505. Epub 2020 Jul 6. PMID 32641236
- [Derived] Guntupalli SR, Brennecke A, Behbakht K, Tayebnejad A, Breed CA, Babayan LM, Cheng G, Ramzan AA, Wheeler LJ, Corr BR, Lefkowits C, Sheeder J, Matsuo K, Flink D. Safety and Efficacy of Apixaban vs Enoxaparin for Preventing Postoperative Venous Thromboembolism in Women Undergoing Surgery for Gynecologic Malignant Neoplasm: A Randomized Clinical Trial. JAMA Netw Open. 2020 Jun 1;3(6):e207410. doi: 10.1001/jamanetworkopen.2020.7410. PMID 32589230

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Apixaban: Oral apixaban 2.5 mg tablet twice daily for 28 days post-surgery
  Oral apixaban: To evaluate the incidence of major bleeding (including clinically relevant non-major (CRNM) bleeding) events in women undergoing surgery for gynecologic cancer with apixaban 2.5 mg twice a day (BID) compared to current standard of care, subcutaneous enoxaparin 40 mg QD for 28 days post surgery.
Period: Overall Study
Arm/Group | Oral Apixaban | Subcutaneous Enoxaparin
Started | 204 | 196
Completed | 204 | 196
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Apixaban | Subcutaneous Enoxaparin | Total
Number analyzed (Participants) | 204 | 196 | 400
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58.0 [21.0 to 87.0] | 58.5 [18.0 to 89.0] | 58.0 [18.0 to 89.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 204 | 196 | 400
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnic group: White Non-Hispanic | 158 | 164 | 322
  Race/ethnic group: Hispanic | 38 | 23 | 61
  Race/ethnic group: African American | 5 | 6 | 11
  Race/ethnic group: Asian | 3 | 3 | 6
Surgical Intervention [Count of Participants; unit: Participants]
  Open | 165 | 152 | 317
  Minimally Invasive | 39 | 44 | 83
Surgeries [Count of Participants; unit: Participants]
  total abdominal hysterectomy(TAH) with BSO/USO | 116 | 112 | 228
  total abdominal hysterectomy (w/out ovaries) | 5 | 3 | 8
  Bilateral/uni salpingo-oophorectomy(BSO)/USO | 42 | 49 | 91
  Radical Hysterectomy | 18 | 24 | 42
  Lymph Node Dissection | 93 | 88 | 181
  Bowel Resection | 25 | 12 | 37
  Removal of Omentum | 82 | 82 | 164
  Surgical Complication | 15 | 10 | 25
Length of Surgery [Median (Inter-Quartile Range); unit: minutes] | 204 [31 to 600] | 215.5 [17 to 743] | 209 [17 to 743]
Confirm Origin [Count of Participants; unit: Participants]
  Uterine Cancer | 65 | 63 | 128
  Ovarian/Fallopian Cancer | 77 | 64 | 141
  Cervical Cancer | 12 | 18 | 30
  Vulva/Vaginal Cancer | 6 | 7 | 13
  Other | 4 | 7 | 11
  Benign | 40 | 37 | 77
Stage [Count of Participants; unit: Participants]
  Low stage (I/II) | 80 | 85 | 165
  High stage (III/IV) | 84 | 74 | 158
  Benign | 40 | 37 | 77
Body-mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 27.4 [11.0 to 50.5] | 26.5 [15.8 to 57.2] | 27.0 [11.0 to 57.2]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Incidence of Major Bleeding
Description: The International Society on Thrombosis and Hemostasis criteria (ISTH) will be used to assess incidence of major bleeding. Participants were monitored for up to 90 days. This is the number of participants who have had at least one major bleeding incidence during the time of observation.
Time Frame: Day 1 post-op/standard of care first medication dose to day 90 (+/-14 days) post-op/standard of care
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Apixaban | Subcutaneous Enoxaparin
Number analyzed (Participants) | 204 | 196
Participants | 1 | 1

2. Primary Outcome: Number of Participants With Incidence of Clinically Relevant Non Major Bleeding Events
Description: Participants were monitored for up to 90 days. This is the number of participants with bleeding events that did not meet the ISTH criteria but still required intervention. This is the number of participants who had at least one non-major bleeding event during the time of observation.
Time Frame: Day 1 post-op/standard of care first dose of medication to day 90 (+/- 14 days) post-op/standard of care
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Apixaban | Subcutaneous Enoxaparin
Number analyzed (Participants) | 204 | 196
Participants | 12 | 19

3. Secondary Outcome: Number of Participants With Incidence of Venous Thromboembolism (VTEs): Deep Vein Thrombosis (DVT) or Pulmonary Embolism (PE)
Description: Participants were monitored for up to 90 days. Both DVTs and PEs will be measured using the Wells criteria, ultrasound, and/or CT. This is the number of participants who had at least one DVT or PE during the time of observation.
Time Frame: Day 1 post-op/standard of care to day first dose of medication 90 (+/- 14 days) post-op/standard of care
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Apixaban | Subcutaneous Enoxaparin
Number analyzed (Participants) | 204 | 196
Participants | 2 | 3

4. Secondary Outcome: Number of Participants Who Met Medication Adherence Rates
Description: Participants were monitored for up to 28 days. This was measured through self-report, patient diaries, and the return of all medication bottles/syringes. This was the number of participants that did not miss more than 2 days of study medication over 28 days (less than 4 pills or 2 injections missed).
Time Frame: Day 1 post-op/standard of care first dose of medication to Day 28 (+/- 4 days) post-op/standard of care
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Apixaban | Subcutaneous Enoxaparin
Number analyzed (Participants) | 204 | 196
Participants | 173 | 164

5. Secondary Outcome: Number of Participants With a Patient Satisfaction Assessment
Description: Participants were monitored at the 28 (+/- 4) day post-op visit. This was measured through administering a participant satisfaction questionnaire ranging from strongly agree to strongly disagree.This is the number of participants that completed the questionnaire in response to agreeing it was difficult to remember to take the medication, agreeing that there was pain associated with the medication, and agreeing that the medication was easy to use.
Time Frame: On visit 4, which is 28 days (+/- 4 days) post-op/standard of care
Population: One patient did not answer the "pain associated with taking the medication" category.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Apixaban | Subcutaneous Enoxaparin
Number analyzed (Participants) | 188 | 187
Participants
  Difficult remembering to take medication: Agree | 23 | 23
  Difficult remembering to take medication: Neutral | 16 | 15
  Difficult remembering to take medication: Disagree | 149 | 149
  Pain associated with taking the medication: number analyzed (Participants) | 187 | 187
  Pain associated with taking the medication: Agree | 4 | 92
  Pain associated with taking the medication: Neutral | 10 | 25
  Pain associated with taking the medication: Disagree | 173 | 70
  Was medication easy to take: Agree | 186 | 110
  Was medication easy to take: Neutral | 2 | 21
  Was medication easy to take: Disagree | 0 | 56

6. Secondary Outcome: Change in Quality of Life From Baseline to 28 Days Post-op
Description: This was measured through a validated health survey (SF-8™) provided by a healthcare company (Optum®), which measured overall physical and mental well-being, with responses ranging from none to very, not at all to extremely, etc. Change was calculated as the difference at baseline versus 28 days post op. The score was 0-100 and a higher score was considered a better outcome.
Time Frame: At baseline, and visit 4, which is 28 days (+/- 4 days) post-op/standard of care
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Oral Apixaban | Subcutaneous Enoxaparin
Number analyzed (Participants) | 204 | 196
score on a scale
  physical score-baseline | 50.7 [19.2 to 64.5] | 49.7 [16.2 to 62.7]
  physical score-visit 4 | 39.2 [21.0 to 58.6] | 38.5 [17.8 to 60.7]
  Physical change | -5.9 [-35.4 to 30.5] | -6.2 [-36.1 to 28.7]
  mental score-baseline | 50.7 [19.2 to 64.5] | 49.7 [16.2 to 62.7]
  mental score-visit 4 | 50.7 [18.5 to 69.4] | 49.3 [19.7 to 62.2]
  Mental change | 0.8 [-30.3 to 30.8] | 0.0 [-30.7 to 41.1]

ADVERSE EVENTS:
Time Frame: 90 (+/- 14) days post first study medication dose
Arm/Group | Oral Apixaban | Subcutaneous Enoxaparin
All-Cause Mortality (participants affected / at risk) | 2/204 | 2/196
Serious Adverse Events (participants affected / at risk) | 13/204 | 14/196
Other Adverse Events (participants affected / at risk) | 53/204 | 45/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Apixaban (N=204) | Subcutaneous Enoxaparin (N=196)
Admitted for abdominal pain and emesis (Gastrointestinal disorders) | 0 | 1
Admitted for ileus (Surgical and medical procedures) | 1 | 0
Admitted for wound Infection (Surgical and medical procedures) | 1 | 3
Admitted for neutropenic fever from chemotherapy (General disorders) | 1 | 1
Admitted for pneumonia (General disorders) | 0 | 2
Admitted for excess kidney fluid and stent placement (General disorders) | 0 | 1
Admitted for Nausea/emesis from chemotherapy (General disorders) | 3 | 0
Admitted for dehydration (General disorders) | 2 | 2
Admitted for clostridium difficile (Gastrointestinal disorders) | 0 | 1
Admitted for small bowel obstruction (General disorders) | 1 | 2
Admitted for pelvic infection (General disorders) | 1 | 0
Admitted for wound closure (General disorders) | 0 | 1
Admitted for vaginal cuff bleeding from open vessel from surgery stitches (Surgical and medical procedures) | 1 | 0
Admitted for nausea and stomach flu (General disorders) | 1 | 0
Admitted for ongoing UTI/sepsis - resolved (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Apixaban (N=204) | Subcutaneous Enoxaparin (N=196)
Hematoma (Blood and lymphatic system disorders) | 1 | 5
Wound infection (Surgical and medical procedures) | 7 | 10
Dizziness (General disorders) | 10 | 1
Suspected allergic reaction (General disorders) | 1 | 1
Arthralgia (General disorders) | 7 | 2
Bruising (General disorders) | 4 | 11
Skin rash/cellulitis (General disorders) | 1 | 2
Vaginal spotting/discharge/bleeding (General disorders) | 4 | 1
Epistaxis (General disorders) | 3 | 2
Abscess/discharge from incision (General disorders) | 2 | 0
Headache (General disorders) | 7 | 5
Hospitalized in 28 days (General disorders) | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/71/NCT02366871/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2020-01-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT02366871/Prot_SAP_001.pdf